CLINICAL TRIAL: NCT04912388
Title: Serum Cytokine Levels in Patients with Lumbal Disc Herniation with and Without Neurological Deficits and Effectiveness of Exercise
Brief Title: Serum Cytokine Levels in Patients with Lumbal Disc Herniation and Effectiveness of Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, birgül morkoç, Principal investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KA-20040
Record Dates: First submitted 2021-05-28; First posted 2021-06-03 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-03

CONDITIONS: Low Back Pain
Keywords: Low back pain; Disc herniation; Stabilization exercises; General exercises; Cytokines; Inflammation
MeSH Terms: conditions — Low Back Pain; Intervertebral Disc Displacement; Inflammation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- The stabilization group (Experimental): The stabilization group will perform lumbal stabilization exercises in lying, sitting, standing and on a swisball 3 times a week during 6 weeks.
  Interventions: Other: Lumbal stabilization excercises
- The general exercise group (Experimental): The general exercise group will perform conventional exercises 3 times a week during 6 weeks.
  Interventions: Other: Conventional exercises
- The control group (No Intervention): Individuals in the control group will not be treated.

INTERVENTIONS:
Other: Lumbal stabilization excercises — The stabilization group will perform lumbal stabilization exercises in lying, sitting, standing and on a swisball 3 times a week during 6 weeks.
  Arms: The stabilization group
Other: Conventional exercises — The general exercise group will perform conventional exercises 3 times a week during 6 weeks.
  Arms: The general exercise group

SUMMARY:
The aim of the study is to investigate serum cytokine levels and the efficacy of lumbar stabilization exercises in patients with lumbar disc herniation with and without neurological deficits. Patients who applied to Hacettepe University Hospitals Physical Medicine and Rehabilitation Department with low back pain complaints and were referred for treatment will be included in the study.

DETAILED DESCRIPTION:
The aim of the study is to investigate serum cytokine levels and the efficacy of lumbar stabilization exercises in patients with lumbar disc herniation with and without neurological deficits. Patients who applied to Hacettepe University Hospitals Physical Medicine and Rehabilitation Department with low back pain complaints and were referred for treatment will be included in the study. Healthy individuals of similar age, height and weight will also be included for references to normal serum cytokine levels. All patients will be evaluated twice, before and 6 weeks after treatment. The treatment program will be applied 3 times a week for 6 weeks under the supervision of a physiotherapist.

ELIGIBILITY:
Inclusion Criteria for patients with disc herniation:

* Diagnosis of disc herniation (protrusion, extrusion, sequestered disc)
* not an indication for lumbar disc herniation surgery
* for patients with neurological deficits, loss of strength, decrease in DTRs, loss of sensation and at least one positive SLR test and presence of radicular pain
* pain intensity of VAS ≥ 3
* male and female patients between the ages of 20-55

Inclusion Criteria for heathy people

* not having low back pain complaints in the past
* female and male healthy individuals between the ages of 20-55

Exclusion Criteria:

* systemic or inflammatory disease
* pregnant or breastfeeding women
* surgery of lumbar region
* fracture of lumbar vertebrae
* lumbar scoliosis
* medication use for psychiatric disorders
* tumor
* allergy
* neurological disease
* alcohol-drug use
* generalized musculoskeletal pain

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 111 (Actual)
Dates: Start 2021-07-30 (Actual); Primary Completion 2024-02-23 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
inflammatory cytokines | 6 weeks
  Tnf-alfa , IL-6, IL-4, IL-1β, Beta-endorphins, Anandamide, Arachidonoylgylycerol will be evaluated with ELISA kit.

CONTACTS AND LOCATIONS:
Overall Officials: Birgül Morkoç, PhD student, Principal Investigator — Hacettepe University
Locations (1):
- Faculty of Physiotherapy and rehabilitation, Ankara, Altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Non are planned to be shared